CLINICAL TRIAL: NCT00006349
Title: An Exploratory Trial of Donepezil and Vitamin E to Prevent Cognitive Dysfunction in Patients With Small Cell Lung Cancer (SCLC) After Cancer Treatment Which Includes Prophylatic Cranial Irradiation (PCI)
Brief Title: Donepezil and Vitamin E to Prevent Side Effects Caused By Radiation Therapy to the Head in Patients Receiving Treatment for Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N99C5; CDR0000068206 (Registry Identifier: PDQ (Physician Data Query)); NCI-P00-0169
Record Dates: First submitted 2000-10-04; First posted 2003-05-29 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cognitive/Functional Effects; Delirium; Depression; Lung Cancer; Radiation Toxicity
Keywords: depression; delirium; cognitive/functional effects; radiation toxicity; limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Delirium; Depression; Lung Neoplasms; Radiation Injuries; Small Cell Lung Carcinoma | interventions — Vitamin E; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- donepezil + vitamin E (Experimental): Patients receive oral donepezil daily and vitamin E twice daily.
  All patients begin treatment within 2 weeks after completion of prophylactic cranial irradiation. Treatment continues for a minimum of 1 month in the absence of disease progression, unacceptable toxicity, or a 3.0 point drop on the Mini Mental State Examination (MMSE) and/or a 5 point drop on the Blessed Dementia Scale.
  Cognition is assessed using the Blessed Dementia Scale and the MMSE at baseline and then every 3 months during study.
  Quality of life and depression are assessed at baseline and then every 3 months during study.
  Patients are followed every 6 months.
  Interventions: Dietary Supplement: vitamin E; Drug: donepezil hydrochloride
- placebo (Placebo Comparator): Patients receive oral placebo twice daily.
  All patients begin treatment within 2 weeks after completion of prophylactic cranial irradiation. Treatment continues for a minimum of 1 month in the absence of disease progression, unacceptable toxicity, or a 3.0 point drop on the Mini Mental State Examination (MMSE) and/or a 5 point drop on the Blessed Dementia Scale.
  Cognition is assessed using the Blessed Dementia Scale and the MMSE at baseline and then every 3 months during study.
  Quality of life and depression are assessed at baseline and then every 3 months during study.
  Patients are followed every 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: vitamin E
  Arms: donepezil + vitamin E
Drug: donepezil hydrochloride
  Arms: donepezil + vitamin E
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Donepezil and vitamin E may be able to decrease side effects caused by radiation therapy given to prevent brain metastases in patients with small cell lung cancer. It is not yet known if donepezil and vitamin E are effective in preventing side effects caused by radiation therapy to the head.

PURPOSE: Randomized phase III trial to determine the effectiveness of donepezil and vitamin E in preventing side effects caused by radiation therapy given to prevent brain metastases in patients who have small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the interval between completion of cancer treatment that included prophylactic cranial irradiation and onset of cognitive decline in patients with small cell lung cancer (SCLC) treated with donepezil and vitamin E vs placebo.
* Determine the toxicity of donepezil and vitamin E in these patients.
* Determine whether preserved cognitive function favorably impacts quality of life in these patients.
* Determine the natural history of cognitive decline in these patients after cancer treatment.
* Determine whether genotypes of apolipoprotein E predict decline in cognitive function among patients at risk for treatment-associated dementia and whether these genotypes predict duration of disease-free survival among patients who have achieved complete response after treatment for SCLC.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to cognitive function (normal vs mild to moderate dysfunction vs severe dysfunction) and age (60 and under vs over 60).

Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral donepezil daily and vitamin E twice daily.
* Arm II: Patients receive oral placebos according to the same schedule as the study drugs in arm I.

All patients begin treatment within 2 weeks after completion of prophylactic cranial irradiation. Treatment continues for a minimum of 1 month in the absence of disease progression, unacceptable toxicity, or a 3.0 point drop on the Mini Mental State Examination (MMSE) and/or a 5 point drop on the Blessed Dementia Scale.

Cognition is assessed using the Blessed Dementia Scale and the MMSE at baseline and then every 3 months during study.

Quality of life and depression are assessed at baseline and then every 3 months during study.

Patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of small cell lung cancer (SCLC)

  * Must meet one of the following conditions:

    * Enrolled no more than 4 weeks before initiation of prophylactic cranial irradiation (PCI) OR
    * Enrolled no more than 10 days after initiation of PCI
  * Limited or extensive stage SCLC with complete response (CR) outside chest allowed
* Must have CR or minimal disease after completion of intended course of chemotherapy
* No disease progression since initiation of PCI
* No prior or concurrent CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 2 times upper limit of normal

Cardiovascular:

* No sick sinus syndrome or other symptomatic supraventricular conduction disorders even if symptoms currently controlled by antiarrhythmics

Pulmonary:

* No history of asthma or chronic obstructive pulmonary disease requiring chronic oxygen therapy

Other:

* No medical or psychiatric condition that would increase risk
* No seizure disorder
* No ongoing alcohol abuse

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* See Disease Characteristics
* No concurrent anticancer chemotherapy

Other:

* No concurrent medications that would impair baseline cognitive function or are likely to be dose escalated over the next few months
* No other concurrent vitamin E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2001-02; Primary Completion 2005-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Compare the interval between completion of cancer treatment that included prophylactic cranial irradiation and onset of cognitive decline in patients with small cell lung cancer (SCLC) treated with donepezil and vitamin E vs placebo | Up to 6 months

SECONDARY OUTCOMES:
Quality of life | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (15):
- United States (15):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jatoi A, Kahanic SP, Frytak S, Schaefer P, Foote RL, Sloan J, Petersen RC. Donepezil and vitamin E for preventing cognitive dysfunction in small cell lung cancer patients: preliminary results and suggestions for future study designs. Support Care Cancer. 2005 Jan;13(1):66-9. doi: 10.1007/s00520-004-0696-0. Epub 2004 Oct 9. PMID 15480814